CLINICAL TRIAL: NCT04947839
Title: Novel Equation for Estimating Resting Energy Expenditure in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor in Renal Division，Department of Medicine, Peking University First Hospital
Other Study IDs: REE equation in dialysis
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Resting Energy Expenditure; Peritoneal Dialysis; Equation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The energy and nutrition states are closely associated with dialysis patients' complications and outcomes. To reach the energy balance target, we need the accurate resting energy expenditure level of patients. Traditional equations do not focus on and applicable to peritoneal dialysis patients, so we aim to develop and validate an equation for estimating resting energy expenditure in peritoneal patients.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients and hemodialysis patients
* Dialysis length >3 months
* >18 years old
* Consented to participate in all aspects of the study

Exclusion Criteria:

* Acute complications to hospitalization 1 month prior to the study;
* Acute or chronic infections, cancer, and other wasting diseases in the past year;
* Thyroid dysfunction;
* Acute onset of podagra; Musculoskeletal diseases;
* Respiratory diseases (asthma, pleural effusion, pneumothorax, COPD);
* History of hormonal drug use;
* During pregnancy or lactation;
* Can not maintain posture and complete the REE test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All peritoneal dialysis patients meet the inclusion and exclusion criteria in a single center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Novel equation development | March 18, 2021 to October 30, 2021
  Developed equation for estimating resting energy expenditure in peritoneal dialysis patients
Novel equation validation | October 30, 2021 to December 30, 2021
  Validate the novel equation with resting energy expenditure obtained by indirect calorimetry (IC).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Haidian Hospital, Beijing